CLINICAL TRIAL: NCT02062151
Title: Acupuncture Use in Infants Treated for Neonatal Abstinence Syndrome: a Pilot Study
Brief Title: Acupuncture in Neonatal Abstinence Syndrome (NAS) Babies
Acronym: AA NAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Acupuncture for NAS
Record Dates: First submitted 2014-02-05; First posted 2014-02-13 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: Acupuncture
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NAS babies (Experimental): Acupuncture for NAS
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture

SUMMARY:
This pilot study is intended to assess feasibility of auricular acupuncture in NAS infants who require pharmacologic therapy. We intend to evaluate acceptability of auricular acupuncture, infant tolerance, recruitment strategies, and methodological issues. We plan to also test and generate hypotheses in preparation to apply for funding a larger randomized controlled trial.

DETAILED DESCRIPTION:
Objectives:

Primary: To establish feasibility of a protocol for auricular acupuncture in infants suffering from NAS admitted to the NICU receiving pharmacologic therapy.

Secondary: In infants suffering from NAS admitted to the Neonatal Intensive Care Unit (NICU) receiving pharmacologic therapy:

1. Determine parent and staff acceptability of auricular acupuncture
2. Determine infant tolerance to auricular acupuncture
3. Evaluate the effect of auricular acupuncture on individual items of the Modified Finnegan Neonatal Abstinence Severity score associated with sympathetic nervous system responses
4. Evaluate the effect of auricular acupuncture on time to return to birth weight

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ≥37.0 wks assessed by the obstetrical team from dating of last menstrual period, ultrasound, or best obstetric estimate
2. Admitted to NICU with diagnosis of NAS requiring pharmacologic therapy
3. Parents give written consent within 72 hours of infant receiving first dose of methadone

Exclusion Criteria:

1. Helix or antihelix of ear is deformed and needle is unable to be placed
2. A suspected or confirmed genetic or metabolic syndrome
3. Custody retained by the Department of Children and Families
4. Any skin condition involving the ear(s)
5. Suspected or documented infection at the time of enrollment

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Weathers, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NAS Babies
Started | 21
Completed | 20
Not Completed | 1
Not completed — screen failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | NAS Babies
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 20
duration of nicu admission [Mean (Standard Deviation); unit: days] | 26 (15)
duration of methadone treatment [Mean (Standard Deviation); unit: days] | 21 (14)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Skin Breakdown and / or Cellulitis
Time Frame: up to 57 days
Measure: Number; unit: participants
Arm/Group | NAS Babies
Number analyzed (Participants) | 20
participants | 0

2. Primary Outcome: Percentage of Dislodged Needles
Time Frame: Within three days of placement
Measure: Number; unit: percentage of needles
Units Other Than Participants: placed needles
Arm/Group | NAS Babies
Number analyzed (Participants) | 20
Number analyzed (placed needles) | 394
percentage of needles | 2

ADVERSE EVENTS:
Groups:
- NAS Babies: Acupuncture for NAS
  Acupuncture
Arm/Group | NAS Babies
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAS Babies (N=20)
MRI with acupuncture needle in place (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes